CLINICAL TRIAL: NCT02594852
Title: Laser - a New Possibility in Fertility Treatment - a Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too few patients enrolling + laser no longer available
Sponsor: Regionshospitalet Viborg, Skive (Other)
Responsible Party: Principal Investigator, Helle Olesen Elbaek, Clinical Director, M.D, Regionshospitalet Viborg, Skive
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-288-14
Record Dates: First submitted 2015-05-28; First posted 2015-11-03 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Infertility; Exposure Laser
MeSH Terms: conditions — Infertility | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (+ laser) (Experimental): + laser therapy
  Interventions: Device: + laser
- Non-intervention (- laser) (Placebo Comparator): - laser
  Interventions: Device: + laser

INTERVENTIONS:
Device: + laser — Use of laser in the treatment

SUMMARY:
In this study the investigators want to investigate if the pregnancy rate in conjunction with fertility treatment increases with concomitant use of laser therapy.

DETAILED DESCRIPTION:
Furthermore the investigators want to examine the participants general mental and physical wellbeing during the experimental period using a VAS-scale.

ELIGIBILITY:
Inclusion Criteria:

1. BMI : 18-32
2. long agonist/short antagonist IVF/intracytoplasmatic sperm injection (ICSI)treatment
3. 1-2 IVF/ICSI treatments without obtaining pregnancy.
4. signed consent

Exclusion Criteria:

1. uterine malformations
2. Uterine fibroids/polyps
3. need of an interpreter.
4. D.M, epilepsy, liver-kidney-heart disease
5. endometrial biopsy
6. cancer former cancer disease
7. acupuncture
8. metal in the body
9. suspicious naevi and tatoo´s

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | up to24 months

CONTACTS AND LOCATIONS:
Overall Officials: Helle Elbaek, M.D, Study Director — The Fertility clinic Skive
Locations (1):
- the Fertility clinic, Regional Hospital Skive, Skive, Central Jutland, Denmark